CLINICAL TRIAL: NCT02552485
Title: Prospective, Monocentric Study for the Evaluation of Latent Pulmonary Arterial Hypertension in Patients With Congenital Shunt Lesions Lost to Follow-up.
Brief Title: Evaluation of Latent Pulmonary Arterial Hypertension in Congenital Shunt Lesions
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, prof. dr. Werner Budts, Prof. dr. Werner Budts, Universitaire Ziekenhuizen KU Leuven
Other Study IDs: S56867
Record Dates: First submitted 2015-09-10; First posted 2015-09-17 (Estimated); Last update posted 2015-12-31 (Estimated); Status verified 2015-12

CONDITIONS: Atrial Septal Defects; Ventricular Septal Defects
MeSH Terms: conditions — Heart Septal Defects, Atrial; Heart Septal Defects, Ventricular

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: No intervention was applied, because it is an observational study

SUMMARY:
Prospective, monocentric study for the evaluation of latent pulmonary arterial hypertension in patients with congenital shunt lesions lost to follow-up. Lost to follow-up is defined as latest clinical control ≥ 5 years.

DETAILED DESCRIPTION:
Pulmonary arterial hypertension (PAH) in patients with congenital heart disease (CHD) usually develops secondary to chronic volume overload of the pulmonary circulation following left to right shunt. This overload leads to elevated pulmonary artery pressure (PAP) and later to increased pulmonary vascular resistance (PVR). This causes pressure overload in the right heart, and thereby right ventricular (RV) and right atrial (RA) dysfunction, which may implicate considerable morbidity and even mortality. Since PAH nowadays is mostly detected when symptoms occur and PAP are elevated, the disease already evolved to an advanced (partially irreversible) stage and treatment is often initiated too late.

Dismissal from follow-up after a surgical correction of simple CHD was customized in the seventies and eighties. There is no literature available that learns us whether these patients really need follow-up or not. A substantial number must have insidiously developed PAH or mild pulmonary vascular disease (PVD) and still are prone to develop PAH later in life. It is relevant to recall these patients dismissed from follow-up in the past, because they might carry a lot of useful information on the natural history of PAH development. Focus will lie mainly on patients with simple shunt lesions, as atrial septal defect (ASD) and ventricular septal defect (VSD).

ELIGIBILITY:
Inclusion Criteria:

* Previous repair for secundum ASD, VSD

Exclusion Criteria:

* Other congenital heart disease
* Chronic lung disease or total lung capacity < 80% of predicted value
* History of pulmonary embolism

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent congenital heart defect closure before the age of 18 years and who are lost to follow-up. Lost to follow-up is defined as latest clinical control ≥ 5 years.
Sampling Method: Probability Sample
Enrollment: 93 (Actual)
Dates: Start 2015-01; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Mortality | From date of birth until date of study inclusion (up to 100 months)

CONTACTS AND LOCATIONS:
Overall Officials: Werner Budts, MD, PhD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- UZLeuven, Leuven, Belgium